CLINICAL TRIAL: NCT05697380
Title: Communication Bridge: A Person-centered Internet-based Intervention for Individuals With Primary Progressive Aphasia 3.0 Pilot
Brief Title: CB3 Pilot (Communication Bridge: A Person-centered Internet-based Intervention for Individuals With Primary Progressive Aphasia)
Acronym: CB3 Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-1333; 2R56AG055425-06 (NIH); R01AG055425 (NIH)
Record Dates: First submitted 2023-01-10; First posted 2023-01-25 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Aphasia; Primary Progressive Aphasia; Dementia; Communication; Alzheimer Disease
MeSH Terms: conditions — Aphasia; Aphasia, Primary Progressive; Dementia; Communication; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Communication Bridge™ (Experimental): Participants receive Communication Bridge™, a multi-component, participation-focused, dyadic intervention in which both the person with PPA and their co-enrolled communication partner are intervention recipients. Communication Bridge™ is modelled on the Living with Aphasia: Framework for Outcome Measurement (A-FROM) and the Care Pathway Model that was developed for persons living with primary progressive aphasia. Consistent with participation-focused intervention models personally salient training stimuli are incorporated into all therapy activities in the Experimental arm.
  Interventions: Behavioral: Communication Bridge™

INTERVENTIONS:
Behavioral: Communication Bridge™ — Evidence-based speech language therapy treatment will be compared and contrasted.

SUMMARY:
This study will evaluate evidence-based treatments for adults with mild Primary Progressive Aphasia (PPA). The aim of the study is to help identify efficacious communication and quality of life interventions for those with PPA and their care-partners.

Participants with a diagnosis of PPA and their actively-engaged care partners will be involved in the study for 12 months. Each participant will receive a iPad equipped with the necessary applications and features for the study. Participants will complete evaluations, speech therapy sessions with a speech and language therapist, and sessions with a licensed social worker or related clinician. They will have access to Communication Bridge, a personalized web application to practice home exercises that reinforce treatment strategies. There are no costs to participate in this study.

DETAILED DESCRIPTION:
This study will evaluate evidence-based treatments for adults with mild Primary Progressive Aphasia (PPA). The aim of the study is to help identify efficacious communication and quality of life interventions for those with PPA and their care-partners.

Participants with a diagnosis of PPA and their actively-engaged care partners will be involved in the study for 12 months. Each participant will receive a iPad equipped with the necessary applications and features for the study. Participants will complete evaluations, speech therapy sessions with a speech and language therapist, and sessions with a licensed social worker or related clinician. They will have access to Communication Bridge, a personalized web application to practice home exercises that reinforce treatment strategies. There are no costs to participate in this study.

ELIGIBILITY:
Inclusion Criteria (person with PPA):

1. Meets diagnostic criteria for PPA based on neurologist and supporting medical assessments (extracted from medical records)
2. English as primary language used in daily communication activities (by self-report)
3. Adequate hearing (aided or unaided) for communicating with others in a crowded room (by self-report)
4. Adequate vision (aided or unaided) for reading a newspaper, or other functional materials (by self-report)
5. Able to pass technology screening and demonstrates sufficient knowledge for use of video conference and Communication Bridge™ web application use (with or without training)

Exclusion Criteria:

* A dementia diagnosis other than Primary Progressive Aphasia
* Participation is co-enrolled in an outside speech language therapy program during the study course.
* Communication partners will be excluded if they have a pre-existing communication impairment that would affect study participation (e.g., aphasia, dementia) Medical records may be requested and reviewed to determine eligibility.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Healthy Aging & Alzheimer's Research Care Center (University of Chicago), Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Communication Bridge™ (PPA Participants); Experimental: Communication Bridge™ (Care Partners): Participants receive Communication Bridge™, a multi-component, participation-focused, dyadic intervention in which both the person with PPA and their co-enrolled communication partner are intervention recipients. Communication Bridge™ is modelled on the Living with Aphasia: Framework for Outcome Measurement (A-FROM) and the Care Pathway Model that was developed for persons living with primary progressive aphasia. Consistent with participation-focused intervention models personally salient training stimuli are incorporated into all therapy activities in the Experimental arm.
  Communication Bridge™: Evidence-based speech language therapy treatment will be compared and contrasted.
Period: Overall Study
Arm/Group | Experimental: Communication Bridge™ (PPA Participants) | Experimental: Communication Bridge™ (Care Partners)
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Communication Bridge™ (Care-Partners): Participants receive Communication Bridge™, a multi-component, participation-focused, dyadic intervention in which both the person with PPA and their co-enrolled communication partner are intervention recipients. Communication Bridge™ is modelled on the Living with Aphasia: Framework for Outcome Measurement (A-FROM) and the Care Pathway Model that was developed for persons living with primary progressive aphasia. Consistent with participation-focused intervention models personally salient training stimuli are incorporated into all therapy activities in the Experimental arm.
  Communication Bridge™: Evidence-based speech language therapy treatment will be compared and contrasted.
- Total: Total of all reporting groups
Arm/Group | Experimental: Communication Bridge™ (PPA Participants) | Experimental: Communication Bridge™ (Care-Partners) | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Highest Degree Earned [Count of Participants; unit: Participants]
  Did not complete high school | 0 | 0 | 0
  High School/GED | 0 | 1 | 1
  Some College | 0 | 2 | 2
  Bachelor's Degree | 3 | 0 | 3
  Master's Degree | 1 | 1 | 2
  Advanced Graduate/Phd | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Communication Confidence (CCRSA)
Description: Communication Confidence Rating Scale in Aphasia, a 0-100 numeric rating scale with 0 representing 'not confident' and 100 representing 'very confident'. Higher scores indicate greater confidence. (Note Primary Outcome Measure was not collected for care-partners)
Time Frame: Time Frame: 5 assessment time points through study completion, an average of 1 year, including change over time
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Communication Bridge™ (PPA Participants)
Number analyzed (Participants) | 4
score on a scale
  Block 4 Evaluation (Baseline) | 64.32 (8.60)
  Post-Intervention Evaluation 4 (at 2 months) | 65.91 (6.90)
  Block 5 Evaluation (at 6 months) | 63.00 (8.31)
  Post-Intervention Evaluation 5 (at 8 months) | 64.77 (9.72)
  Block 6 Evaluation (at 12 months) | 61.36 (12.19)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of 1 year from the participant's enrollment at baseline.
Description: Adverse Event Reporting below if for the PPA Participant Group ONLY.
Arm/Group | Experimental: Communication Bridge™ (PPA Participants) | Experimental: Communication Bridge™ (Care Partners)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Communication Bridge™ (PPA Participants) (N=4) | Experimental: Communication Bridge™ (Care Partners) (N=4)
Medical Event (Surgical and medical procedures) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Communication Bridge™ (PPA Participants) (N=4) | Experimental: Communication Bridge™ (Care Partners) (N=4)
Other psychosocial events (Psychiatric disorders) | 0 (0) | 2 (2)
medical event (non serious) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT05697380/Prot_000.pdf